CLINICAL TRIAL: NCT00786929
Title: Randomized Controlled Trial on Sterile Fluid Collections Management in Acute Pancreatitis
Brief Title: Acute Pancreatitis and Acute Fluid Collections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center, Tuzla (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MB-68/02
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2008-11

CONDITIONS: Pancreatitis
Keywords: Conversion to more aggressive treatment of recurrent fluid collection
MeSH Terms: conditions — Pancreatitis | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- drainage (Experimental)
  Interventions: Procedure: Catheter drainage
- 2 (Active Comparator): Conservative treatment
  Interventions: Drug: Conservative treatment

INTERVENTIONS:
Procedure: Catheter drainage
  Arms: drainage
Drug: Conservative treatment
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate if percutaneous drainage of sterile fluid collections recurring after initial aspiration in acute pancreatitis yielded better results than their conservative management.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and signs of acute pancreatitis and if pancreatic or/and peripancreatic fluid collections were confirmed by ultrasound and computed tomography examination

Exclusion Criteria:

* Collections resulting from pancreatic surgery, chronic pancreatitis and encapsulated collections and collections with uncertainty about the relationship between the collections and clinical symptoms and signs of acute pancreatitis were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2003-03; Primary Completion 2007-02 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Conversion to more aggressive procedure | Sep 2007

SECONDARY OUTCOMES:
Number of patients turning culture positive, length of hospital stay, catheter dwell time, catheter problems and changes per patient | Oct 2007

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Center, Tuzla, TK, Bosnia and Herzegovina

REFERENCES:
- [Background] Bradley EL 3rd. A clinically based classification system for acute pancreatitis. Ann Chir. 1993;47(6):537-41. No abstract available. PMID 8105746
- See also: Related Info — http://mc.manuscriptcentral.com/surgendosc
- See also: Related Info — http://ees.elsevier.com/jvir/